CLINICAL TRIAL: NCT05181709
Title: A Phase-1, Open-Label, Placebo-Controlled Evaluation of a Live, Recombinant Newcastle Disease Virus Expressing the Spike Protein of SARS-CoV-2 (NDV-HXP-S), an Investigational Product for Intranasal (IN) and/or Intramuscular (IM) Vaccination in Healthy Adults Previously Immunized Against COVID-19.
Brief Title: A Live Recombinant Newcastle Disease Virus-vectored COVID-19 Vaccine Phase 1 Study.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sean Liu (Other)
Responsible Party: Sponsor-Investigator, Sean Liu, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: STUDY-21-01589
Record Dates: First submitted 2022-01-04; First posted 2022-01-06 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: SARS-CoV-2
Keywords: SARS-CoV-2; COVID-19; Vaccine; Booster
MeSH Terms: conditions — COVID-19 | interventions — Sodium Chloride; NDV-HXP-S COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Random and Sequential Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Cohort 1: Placebo / Sodium Chloride (Placebo Comparator): Participants in Cohort 1 will receive placebo given IN+IM in combination. Placebo administration will be given in an ambulatory setting. IN administration will be immediately followed by IM administration. Participants will be monitored by the research staff for 1-hour after administration. Participants will be permitted to receive any additional federally authorized or approved vaccines 56 days after receiving placebo.
  Interventions: Drug: Sodium Chloride
- Cohort 2: NDV-HXP-S low dose IN (Active Comparator): Participants in Cohort 2 (low, IN) will receive a single administration of a low dose of NDV-HXP-S at 3.3x108 Egg-Infectious Dose50 (EID50). Participants will be given NDV-HXP-S in an ambulatory setting and be monitored by the research staff for 4 hours post-administration. Participants will then return home under home isolation. Home isolation will require daily at-home sample collections and online symptom reporting. Discontinuation of home isolation will require laboratory confirmation of negative NDV-HXP-S virus detection.
  Interventions: Biological: NDV-HXP-S IN low dose
- Cohort 3: NDV-HXP-S low dose IM (Active Comparator): Participants in Cohort 3 (low, IM) will receive a single administration of a low dose of NDV-HXP-S at 3.3x108 Egg-Infectious Dose50 (EID50). Participants will be given NDV-HXP-S in an ambulatory setting and be monitored by the research staff for 4 hours post-administration. Participants will then return home under home isolation. Home isolation will require daily at-home sample collections and online symptom reporting. Discontinuation of home isolation will require laboratory confirmation of negative NDV-HXP-S virus detection.
  Interventions: Biological: NDV-HXP-S IM low dose
- Cohort 4: NDV-HXP-S low dose IN+IM in combination (Active Comparator): Participants in Cohort 4 (low, IN+IM) will receive low doses of NDV-HXP-S at 3.3x108 EID50. Participants will be given NDV-HXP-S in an ambulatory setting where IN and IM doses will be given in succession. Participants will be monitored by the research staff for 4 hours post-administration. Participants will then return home under home isolation. Home isolation will require daily at-home sample collections and online symptom reporting. Discontinuation of home isolation will require laboratory confirmation of negative NDV-HXP-S virus detection.
  Interventions: Biological: NDV-HXP-S IN low dose; Biological: NDV-HXP-S IM low dose
- Cohort 5: NDV-HXP-S high dose IN (Active Comparator): Participants in Cohort 5 (high, IN) will receive high doses of NDV-HXP-S at 1x109 EID50. Participants will ONLY enroll into Cohort 5 if Cohort 2 (low dose IN) did not have any SAEs that required additional participants. Participants will be given NDV-HXP-S in an ambulatory setting and be monitored by the research staff for 4 hours post-administration. Participants will then return home under home isolation. Home isolation will require daily at-home sample collections and online symptom reporting. Discontinuation of home isolation will require laboratory confirmation of negative NDV-HXP-S virus detection.
  Interventions: Biological: NDV-HXP-S IN high dose
- Cohort 6: NDV-HXP-S high dose IM (Active Comparator): Participants in Cohort 6 (high, IM) will receive high doses of NDV-HXP-S at 1x109 EID50. Participants will ONLY enroll into Cohort 6 if Cohort 3 (low dose IM) did not have any SAEs that required additional participants. Participants will be given NDV-HXP-S in an ambulatory setting and be monitored by the research staff for 4 hours post-administration. Participants will then return home under home isolation. Home isolation will require daily at-home sample collections and online symptom reporting. Discontinuation of home isolation will require laboratory confirmation of negative NDV-HXP-S virus detection.
  Interventions: Biological: NDV-HXP-S IM high dose
- Cohort 7: NDV-HXP-S high dose IN+IM in combination (Active Comparator): Participants in Cohort 7 (high, IN+IM) will receive high doses of NDV-HXP-S at 1x109 EID50. Participants will only enroll into Cohort 7 if Cohort 4 did not have an SAE that required additional participants. Participants will be given NDV-HXP-S in an ambulatory setting and be monitored by the research staff for 4 hours post-administration. Participants will then return home under home isolation. Home isolation will require daily at-home sample collection and online symptom reporting. Discontinuation of home isolation will require laboratory confirmation of negative NDV-HXP-S virus detection.
  Interventions: Biological: NDV-HXP-S IN high dose; Biological: NDV-HXP-S IM high dose

INTERVENTIONS:
Drug: Sodium Chloride — Administered intranasal (IN) and intramuscular (IM) in combination
  Other Names: Placebo
  Arms: Cohort 1: Placebo / Sodium Chloride
Biological: NDV-HXP-S IN low dose — Allantoic fluid diluted in Phosphate buffered saline (PBS), to be further diluted to dose strength in sodium chloride.
  Strength: 3.3x108^8 EID50.
  Arms: Cohort 2: NDV-HXP-S low dose IN; Cohort 4: NDV-HXP-S low dose IN+IM in combination
Biological: NDV-HXP-S IM low dose — Allantoic fluid diluted in Phosphate buffered saline (PBS), to be further diluted to dose strength in sodium chloride.
  Strength: 3.3x10^8 EID50.
  Arms: Cohort 3: NDV-HXP-S low dose IM; Cohort 4: NDV-HXP-S low dose IN+IM in combination
Biological: NDV-HXP-S IN high dose — Allantoic fluid diluted in Phosphate buffered saline (PBS). Strength: 1x10^9 EID50.
  Arms: Cohort 5: NDV-HXP-S high dose IN; Cohort 7: NDV-HXP-S high dose IN+IM in combination
Biological: NDV-HXP-S IM high dose — Allantoic fluid diluted in Phosphate buffered saline (PBS). Strength: 1x10^9 EID50.
  Arms: Cohort 6: NDV-HXP-S high dose IM; Cohort 7: NDV-HXP-S high dose IN+IM in combination

SUMMARY:
This study will be a phase-1, open-label, placebo-controlled, evaluation of two-dosages of a live, recombinant Newcastle disease virus expressing the spike protein of SARS-CoV-2 (NDV-HXP-S), an investigational product for IN, IM, or a combined IN+IM vaccination in healthy adults previously immunized against COVID-19. The IN and IM live virus vaccinations will be identical in composition and only differ in route of administration.

DETAILED DESCRIPTION:
Primary Study Objective: To evaluate the safety and tolerability profile of two dose levels of the NDV-HXP-S vaccine as an IN, IM, or a combined administration IN+IM to healthy, previously immunized adults up to 14 days after administration.

Secondary Study Objective: To evaluate the safety and tolerability profile of two dose levels of the NDV-HXP-S vaccine as an IN, IM, or a combined administration IN+IM to healthy, previously immunized adults up to 365 days after administration.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent prior to performing study procedures.
2. Males and non-pregnant females who are between 18 to 59 years of age.
3. Asymptomatic, RT-PCR negative (at screening) AND without a known prior history of COVID-19 infection (requiring a negative SARS-CoV-2 nucleocapsid antibody test result at screening).
4. Provides documentation showing completion of an FDA authorized or approved COVID-19 vaccination regimen, where the last administration was ≥ 6 months (180 days) from the study enrollment date.
5. IF FEMALE PARTICIPANT: A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

   * Is not a woman of child-bearing potential (WOCBP); OR
   * Is a WOCBP and using an acceptable contraceptive method during the intervention period (for a minimum of 90 days after NDV-HXP-S vaccination). The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention. Only highly effective methods of contraception that have a low user dependency or a combination of highly effective methods that are user dependent may be used.
6. IF MALE PARTICIPANT: Agrees to the following requirements during the intervention period and for at least 90 days after NDV-HXP-S vaccination, which corresponds to the time needed to eliminate reproductive safety risk of the study intervention(s):

   * Refrain from donating sperm AND be abstinent from heterosexual intercourse with a female of childbearing potential as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent; OR
   * Must agree to use a male condom when engaging in any activity that allows for passage of ejaculate to another person. In addition to male condom use, a highly effective method of contraception may be considered in WOCBP partners of male participants.
7. Participant understands and agrees to comply with planned study procedures.
8. Participant agrees to not participate in another clinical trial for treatment of COVID-19 or SARS-CoV-2 through Day 365.
9. Participant agrees to not receive any other vaccination (including COVID-19 vaccines) through day 56 of the study.
10. Provides consent for release of information for hospitalization records and other medically attended visits during the study.

Exclusion Criteria:

1. Clinical and/or laboratory evidence indicative of COVID-19 infection.
2. Demonstrates a STRONG COVID-19 positive antibody serology (>12500 AU/ml per chemiluminescent microparticle immunoassay (including AdviseDx SARS-CoV-2 IgG II)) or a NEGATIVE COVID-19 serology on screening against SARS-CoV-2 spike protein.
3. History of hypersensitivity to egg products.
4. History of severe reactions to vaccinations.
5. Potential for prior NDV exposures (i.e., experience as a bird-handler, poultry farmer, or scientist conducting research with NDV).
6. History of an immunocompromising medical condition (such as primary immunodeficiencies, AIDS, or neutropenia).
7. Current or recent use of immunosuppressive medications (i.e., any systemic corticosteroids, chemotherapeutics, immunoglobulin therapies, etc.) based on the assessment of their half-life by the investigator.
8. Any history of HIV, hepatitis C, hepatitis B (by laboratory testing and/or history), Guillain-Barré syndrome, and/or recent receipt of immunoglobulins and/or blood products.
9. Pregnancy or actively breastfeeding.
10. Other medical condition or abnormal laboratory values which may place participant at increased risk for harm due to participation in the study as determined by the investigator.
11. In the opinion of the investigator that it would be unwise to allow the participant to be randomized into the study, including those persons who the investigator would consider as high risk of SARS-CoV-2 exposure, including healthcare workers with direct patient care and laboratory workers who handle SARS-CoV-2.
12. Participants at higher risk of severe COVID-19, as defined by CDC guidance (https://www.cdc.gov/coronavirus/2019-ncov/need-extra-precautions/index.html), where severity of risk and eligibility will be determined by the investigator. This guidance includes details regarding older adults, people with specific medical conditions, and pregnant and recently pregnant people.
13. Participants with fever or signs of acute infection, including symptoms that could indicate SARS-CoV-2 infection.
14. Participants with a history of chronic rhinitis, nasal septal defect, cleft palate, nasal polyps, or other nasal abnormality that might affect vaccine administration.
15. Participants who prepare food in the food industry and childcare workers who have direct contact with children 5 years of age or younger.
16. Participants who have close or household high-risk contacts including but not limited to:

    * Persons more than or equal to 65 years of age
    * Children less than or equal to 5 years of age.
    * Residents of nursing homes.
    * Persons of any age with significant chronic medical conditions as well as immunosuppression or cancer.

    Women who are pregnant, trying to become pregnant, or breastfeeding.
17. Participants who are students, post-doctoral candidates, or trainees of the study site, or are members of the research staff.
18. Participants with a history of myocarditis or pericarditis and individuals with an abnormal troponin or abnormal ECG as determined by the investigator. Participants with a screening 12-lead ECG that shows an average QTc interval >500 msec, complete left bundle branch block, ST-T interval changes suggestive of myocardial ischemia, second- or third-degree AV block, or serious bradyarrhythmias or tachyarrhythmias should be excluded from study participation.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Number of local and systemic reactions | 14 days
  The safety and tolerability profile assessed by the number of local and systemic reactions.

SECONDARY OUTCOMES:
Number of adverse events (AEs) | 365 days
  The safety and tolerability profile assessed by the number of serious adverse events.
Number of serious adverse events (SAEs) | 365 days
  The safety and tolerability profile assessed by the number of serious adverse events.
Number of medically-attended adverse events (MAAEs) | 365 days
  The safety and tolerability profile assessed by the number of medically-attended adverse events (MAAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Sean Liu, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. To achieve aims in the approved proposal.

REFERENCES:
- [Background] Sun W, McCroskery S, Liu WC, Leist SR, Liu Y, Albrecht RA, Slamanig S, Oliva J, Amanat F, Schafer A, Dinnon KH 3rd, Innis BL, Garcia-Sastre A, Krammer F, Baric RS, Palese P. A Newcastle Disease Virus (NDV) Expressing a Membrane-Anchored Spike as a Cost-Effective Inactivated SARS-CoV-2 Vaccine. Vaccines (Basel). 2020 Dec 17;8(4):771. doi: 10.3390/vaccines8040771. PMID 33348607
- [Background] Punnee Pitisuttithum, Viravarn Luvira, Saranath Lawpoolsri, Sant Muangnoicharoen, Supitcha Kamolratanakul, Chaisith Sivakorn, Piengthong Narakorn, Somchaiya Surichan, Sumalee Prangpratanporn, Suttida Puksuriwong, Steven Lamola, Laina D Mercer, Rama Raghunandan, Weina Sun, Yonghong Liu, Juan Manuel Carreño, Rami Scharf, Weerapong Phumratanaprapin, Fatima Amanat, Luc Gagnon, Ching-Lin Hsieh, Ruangchai Kaweepornpoj, Sarwat Khan, Manjari Lal, Stephen McCroskery, Jason McLellan, Ignacio Mena, Marcia Meseck, Benjaluck Phonrat, Yupa Sabmee, Ratsamikorn Singchareon, Stefan Slamanig, Nava Suthepakul, Johnstone Tcheou, Narumon Thantamnu, Sompone Theerasurakarn, Steven Tran, Thanakrit Vilasmongkolchai, Jessica A White, Adolfo Garcia-Sastre, Peter Palese, Florian Krammer, Kittisak Poopipatpol, Ponthip Wirachwong, Richard Hjorth, Bruce L Innis. Safety and Immunogenicity of an Inactivated Recombinant Newcastle Disease Virus Vaccine Expressing SARS-CoV-2 Spike: Interim Results of a Randomised, Placebo-Controlled, Phase 1/2 Trial. medRxiv 2021.09.17.21263758; doi: https://doi.org/10.1101/2021.09.17.21263758
- [Derived] Slamanig S, Lemus N, Lai TY, Singh G, Mishra M, Abdeljawad A, Boza M, Dolange V, Singh G, Lee B, Gonzalez-Dominguez I, Schotsaert M, Krammer F, Palese P, Sun W. A single immunization with intranasal Newcastle disease virus (NDV)-based XBB.1.5 variant vaccine reduces disease and transmission in animals against matched-variant challenge. Vaccine. 2025 Jan 25;45:126586. doi: 10.1016/j.vaccine.2024.126586. Epub 2024 Dec 12. PMID 39667115

DOCUMENTS (1):
  • Informed Consent Form (2023-01-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT05181709/ICF_000.pdf